CLINICAL TRIAL: NCT00907543
Title: Prospective Randomized Phase III Trial Comparing Preoperative Chemoradiation Therapy (Cisplatin, 5-FU and Radiotherapy Followed by Surgery) to Surgery Followed by Postoperative Chemoradiation (Cisplatin, Epirubicin, 5-FU, Radiotherapy) for Esophageal Cancer
Brief Title: Quality of Life in Neoadjuvant Versus Adjuvant Therapy of Esophageal Cancer Treatment Trial
Acronym: QUINTETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Malthaner (Other)
Responsible Party: Sponsor-Investigator, Richard Malthaner, Sponsor-Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-09-025
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Esophageal Neoplasms
Keywords: esophageal carcinoma; chemotherapy; radiation; surgery; randomized clinical trial; Clinical Trial; Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant Treatment (Other): Preoperative chemotherapy/radiotherapy treatment
  Interventions: Other: Preoperative treatment of chemotherapy and radiation
- Adjuvant Treatment (Experimental): Postoperative chemotherapy/radiotherapy treatment
  Interventions: Other: Postoperative treatment of chemotherapy and radiation

INTERVENTIONS:
Other: Preoperative treatment of chemotherapy and radiation — Cisplatin + 5FU with concurrent radiation followed by surgery
  Arms: Neoadjuvant Treatment
Other: Postoperative treatment of chemotherapy and radiation — Surgery followed by cisplatin + 5FU + epirubicin as indicated by pathological stage with extended beam radiation
  Arms: Adjuvant Treatment

SUMMARY:
The purpose of this study is to compare the results of preoperative chemotherapy and radiation followed by surgery to surgery followed by postoperative chemotherapy and radiation for esophageal cancer.

DETAILED DESCRIPTION:
Patients will be randomized to neo-adjuvant or adjuvant treatment. Quality of life questionnaires will be completed every 2 months up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (> 20 cm from the incisors) or gastroesophageal junction are included.
* No distant metastases (M0).
* Patients will be stratified by stage (clinical N0 versus clinical N1), and surgeon.
* Patients with tumours within 3 cm distal spread into gastric cardia as detected by esophagogastroscopy.
* Resectable mediastinal nodes are eligible.
* No prior chemotherapy for this malignancy.
* No prior radiotherapy that would overlap the field(s) treated in this study.
* Patients with other malignancies are eligible only if > 5 years without evidence of disease or completely resected or treated non-melanoma skin cancer.
* Age > 18 years and able to tolerate tri-modality therapy at the discretion of the treating thoracic surgeon, medical and radiation oncologists. Tumours must be resectable after assessment by the thoracic surgeon.

Exclusion Criteria:

* Cancers of the cervical esophagus (< 20 cm are excluded).
* Tumours that have > 3 cm of spread into cardia of the stomach are considered gastric cancers and are ineligible.
* Patients with biopsy (by endoscopic ultrasound, laparoscopy, or laparotomy ) proven metastatic supraclavicular nodes are ineligible.
* Patients with biopsy proven metastatic celiac nodes are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life as assessed by FACT-E | 1 year

SECONDARY OUTCOMES:
Safety and morbidity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Malthaner, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Malthaner RA, Yu E, Sanatani M, Lewis D, Warner A, Dar AR, Yaremko BP, Bierer J, Palma DA, Fortin D, Inculet RI, Frechette E, Raphael J, Gaede S, Kuruvilla S, Younus J, Vincent MD, Rodrigues GB. The quality of life in neoadjuvant versus adjuvant therapy of esophageal cancer treatment trial (QUINTETT): Randomized parallel clinical superiority trial. Thorac Cancer. 2022 Jul;13(13):1898-1915. doi: 10.1111/1759-7714.14433. Epub 2022 May 24. PMID 35611396